CLINICAL TRIAL: NCT01249014
Title: Study Using Fluid Warming and Forced Air Warming Immediately Prior to and During Elective Cesarean Section
Brief Title: Temperature Study in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward Riley, Principle Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SU-11102010-7189
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Cesarean Section; Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No peri-operative warming.
- Warmed fluids (Experimental): Patients will receive warmed i.v. fluids administered pre- and intra-operatively.
  Interventions: Other: Warmed fluids; Device: Belmont fluid warmer
- Warmed fluids and warm air (Experimental): Patients will receive warmed i.v. fluids administered pre- and intra-operatively, and warmed air blown into a blanket covering the body intra-operatively.
  Interventions: Other: Warmed fluids; Other: Fluid warmer and warming blanket; Device: Belmont fluid warmer; Device: Bair hugger warming blanket

INTERVENTIONS:
Other: Warmed fluids — IV fluids warmed by a Belmont fluid warmer
  Arms: Warmed fluids; Warmed fluids and warm air
Other: Fluid warmer and warming blanket — Warm are blown into a Bair hugger warming blanket covering the patient
  Arms: Warmed fluids and warm air
Device: Belmont fluid warmer — Belmont fluid warmer used to warm fluids
  Arms: Warmed fluids; Warmed fluids and warm air
Device: Bair hugger warming blanket — Bair hugger warming blanket laid on body
  Arms: Warmed fluids and warm air

SUMMARY:
During surgery body temperature can decrease which can adversely affect how people recover from surgery. This is a common problem. We aim to reduce the incidence of this drop in body temperature during surgery by testing the effectiveness of warm intravenous fluids that the patients will receive as they are being infused, and of warm air blown into a blanket covering the body. The control group will not have any active warming methods.

Study group 1 will have the intravenous fluid warmer in the pre- and intraoperative period. Study group 2 will have a forced-air warmer in the intra-operative period as well as the fluid warmer in the pre- and intraoperative period. We will also observe the neonates' vital signs following delivery.

DETAILED DESCRIPTION:
Potential participants will be approached by a member of the research team prior to surgery.

Patients will be fully informed of the study by a study investigator, full written informed consent will be obtained. We will recruit healthy ASA 1 and 2 patients undergoing uncomplicated elective cesarean sections. Patients will be randomised into one of three groups.

Control group will have no active warming. Study group 1 will have pre- and intraoperative intravenous fluid warming. Study group 2 will have the same as study group 1 but with additional intraoperative warming air blown into a blanket covering the body.

Temperature measurements will be taken in the pre-op holding area prior to intravenous fluid administration, and thereafter at 15-minute intervals until one hour post-surgery.

At the same time as temperature monitoring the patients will be assessed for shivering (4 point scale) and will be asked their comfort level with regard to their temperature (5 point scale).

We will record vital signs (measured routinely by the pediatricians at cesarean delivery) from the neonate immediately following delivery. Samples of blood will be taken from the placental cord following delivery to measure cord blood gas results.

We will carry out a chart review looking at the success rate of breast feeding (if applicable).

* We are studying the effect of intravenous fluid warming and forced-air warming on your body temperature at the time of your cesarean section.
* Perioperative hypothermia can have adverse affects on your health and recovery following surgery so the aim of this study is to find ways to prevent or reduce the incidence of hypothermia.
* Participants will be randomized into one of three groups. The control group will not receive any perioperative warming. Study group 1 will have intravenous fluids warmed. Study group 2 will be the same as group 1 with the addition of a forced-air warmer in the operating room. Your temperature will be taken in the pre-op holding area prior to intravenous fluid administration, and thereafter at 15-minute intervals until one hour post-surgery. At the time of the temperature measurements we will also assess any shivering you may have and also question you regarding how warm/cold you feel.
* Following delivery of the placenta we will send one blood sample taken from the placental cord to the biochemistry laboratory for analysis of the cord blood gases. The blood sample will not be stored for future studies.
* We will be observing the vital signs of the neonate immediately following delivery.
* We will be carrying out a chart review looking at the success rate of breast feeding (if applicable).

ELIGIBILITY:
Inclusion Criteria:18-40 years. Healthy term (> 37 weeks) pregnant patients undergoing elective cesarean section with spinal anesthesia.

We will not discriminate with regard to ethnic background. ASA 1 and 2 patients scheduled for elective cesarean sections under spinal anesthesia at LPCH.

Exclusion Criteria:Not ASA 1 or 2 Not spinal anesthetic

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
temperature | immediately prior to surgery upto 3hours post spinal anesthetic
  measured every 15 minutes from spinal anesthetic administration

SECONDARY OUTCOMES:
Fetal pH | Post partum

CONTACTS AND LOCATIONS:
Overall Officials: Edward Riley, Study Director — Stanford University; Gill Hilton, Sub-Investigator — Stanford University; Pervez Sultan, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States